CLINICAL TRIAL: NCT06176365
Title: A Phase III, Randomised, Double-blind, Parallel-group, 76-week, Efficacy and Safety Study of Survodutide Administered Subcutaneously Compared With Placebo in Patients With Obesity Disease in Japanese
Brief Title: A Study to Test Whether Survodutide Helps Japanese People Living With Obesity Disease
Acronym: SYNCHRONIZE™JP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1404-0053
Record Dates: First submitted 2023-12-11; First posted 2023-12-19 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — BI 456906

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Survodutide - 3.6 mg (Experimental)
  Interventions: Drug: Survodutide
- Survodutide - 6.0 mg (Experimental)
  Interventions: Drug: Survodutide
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo matching survodutide

INTERVENTIONS:
Drug: Survodutide — once weekly subcutaneous injection
  Other Names: BI 456906
  Arms: Survodutide - 3.6 mg; Survodutide - 6.0 mg
Drug: Placebo matching survodutide — once weekly subcutaneous injection
  Arms: Placebo group

SUMMARY:
This study is open to adults who are at least 18 years old and have

* a body mass index (BMI) of 35 kg/m² or more and at least one health problem related to their weight, or
* a BMI of 27 kg/m² or more and at least two health problems related to their weight.

People who have either type 2 diabetes, high blood pressure, or increased blood lipids can take part in this study. Only people who have previously not managed to lose weight by changing their diet can participate.

The purpose of this study is to find out whether a medicine called survodutide (BI 456906) helps people living with obesity disease to lose weight. Participants are divided into 3 groups by chance, like drawing names from a hat. 2 groups get different doses of survodutide and 1 group gets placebo. Placebo looks like survodutide but does not contain any medicine.

Every participant has a 2 in 3 chance of getting survodutide. Participants inject survodutide or placebo under their skin once a week for about one and a half years. In addition to the study medicine, all participants receive counselling to make changes to their diet and to exercise regularly.

Participants are in the study for about 1 year and 7 months. During this time, it is planned that participants visit the study site up to 14 times and receive 6 phone calls by the site staff.

The doctors check participants' health and take note of any unwanted effects. The participants' body weight is regularly measured. The results are compared between the groups to see whether the treatment works.

ELIGIBILITY:
Inclusion criteria:

1. Male or female, age ≥18 years at the time of signing informed consent
2. Body Mass Index (BMI)

   * ≥35 kg/m² at screening with the presence of at least one obesity-related comorbidities (treated or untreated) according to the Japan Society for the Study of Obesity (JASSO) guideline OR
   * BMI ≥27 kg/m² at screening with the presence of at least two obesity-related comorbidities (treated or untreated) according to the JASSO guideline For all trial patients, at least one co-morbidity should be the following (i)-(iii).

     i. Type 2 diabetes mellitus (T2DM)
     * Diagnosed with T2DM (defined as Glycosylated haemoglobin A1c (HbA1c) ≥6.5% [≥48 mmol/mol]) at least 180 days prior to screening
     * HbA1c ≥6.5% (48 mmol/mol) and <10% (86 mmol/mol) as measured by the central laboratory at screening
     * Currently treated with either: diet and exercise alone or stable treatment (for at least 3 months prior to screening) with metformin, SGLT-2i, acarbose, sulfonylurea, or glitazone as single agent therapy, or up to 3 antihyperglycaemia medications (metformin, SGLT-2i, acarbose, sulfonylurea, or glitazone) according to local label ii. Hypertension iii. Dyslipidaemia
3. History of at least one self-reported unsuccessful dietary effort to lose body weight
4. Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial
5. Woman of childbearing potential (WOCBP) must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria and instructions on the duration of their use will be provided in the patient information.
6. In the investigator's opinion, patients are well-motivated, capable, and willing to:

   * Learn how to self-inject the Investigational medicinal product (IMP), as required for this protocol (persons with physical limitations who are not able to perform the injections must have the assistance of an individual trained to inject the IMP) OR
   * Inject the IMP or accept injection from a designated person
   * Follow study procedures for the duration of the study, including, but not limited to: follow lifestyle advice (for example, dietary restrictions and exercise and exercise plan), maintain a diary, and complete required questionnaires, and handle the IMP as described in the instructions for use (IFU)

Exclusion criteria:

Obesity:

1. Body weight change (self-reported) >5% within 3 months before screening
2. Treatment with any medication for the indication obesity within 3 months before screening
3. Previous or planned (during the trial period) treatment for obesity with surgery or a weight loss device, or prior surgery of the gastrointestinal (GI) tract that could interfere with body weight The following are allowed: (1) liposuction and/or abdominoplasty, if performed >1 year before screening, (2) lap banding, if the band has been removed >1 year before screening, (3) intragastric balloon, if the balloon has been removed >1 year before screening, (4) duodenal-jejunal bypass sleeve, if the sleeve has been removed >1 year before screening, (5) appendectomy, (6) simple hernia repair, or (7) cholecystectomy.
4. Have obesity induced by other endocrinologic disorders (i.e. Cushing Syndrome) or diagnosed monogenetic or syndromic forms of obesity (i.e. melanocortin 4 receptor deficiency, leptin deficiency, or Prader Willi Syndrome)

   Glycaemia:

   For trial patients without T2DM:
5. History of T1DM or T2DM or treatment with glucose lowering agent started within 3 months before screening

   For trial patients with T2DM:
6. History of T1DM
7. Treatment with any medication for the indication of T2DM other than stated in the inclusion criteria within 3 months before screening (i.e. insulin, amylin analogues, GLP-1R agonists, GLP-1R agonist/insulin/GIP combinations, and DPP-4i)
8. New initiation of any other glucose-lowering investigational drug within 3 months prior to screening for this trial

Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2024-01-16 (Actual); Primary Completion 2025-12-03 (Actual); Study Completion 2025-12-03 (Actual)

PRIMARY OUTCOMES:
Percentage change in body weight from baseline to Week 76 | at baseline, at week 76
Achievement of body weight reduction ≥5% (yes/no) from baseline to Week 76 | at baseline, at week 76

SECONDARY OUTCOMES:
Achievement of body weight reduction ≥10% (yes/no) from baseline to Week 76 | at baseline, at week 76
Achievement of body weight reduction ≥15% (yes/no) from baseline to Week 76 | at baseline, at week 76
Achievement of body weight reduction ≥20% (yes/no) from baseline to Week 76 | at baseline, at week 76
Absolute change from baseline to Week 76 in body weight (kg) | at baseline, at week 76
Absolute change from baseline to Week 76 in body mass index (BMI) (kg/m²) | at baseline, at week 76
Absolute change from baseline to Week 76 in waist circumference measured at umbilical level (cm) | at baseline, at week 76
Absolute change from baseline to Week 76 in waist circumference measured at midway between the lower rib margin and the iliac crest (cm) | at baseline, at week 76
Absolute change from baseline to Week 76 in systolic blood pressure (SBP) (mmHg) | at baseline, at week 76
Absolute change from baseline to Week 76 in diastolic blood pressure (DBP) (mmHg) | at baseline, at week 76
Absolute change from baseline to Week 76 in "Capacity to Resist" domain score of the Eating Behaviour Patient reported outcome (PRO) | at baseline, at week 76
  The "Capacity to Resist domain score" of the Eating Behaviour Patient reported outcome (PRO) (units on a scale) will be derived as the sum of items in the domain (possible responses being 0="Not at all", 1="A little", 2="Moderately", 3="A lot", 4="Extremely").
  The domain score is ranging between 0 and 24 and a higher score indicates a lower capacity to resist.
Absolute change from baseline to Week 76 in Eating Behaviour PRO total score | at baseline, at week 76
  The Eating Behaviour PRO total score (units on a scale) will be derived from the "Desire to Eat" and "Capacity to Resist" domain as the sum of all items (possible responses being 0="Not at all", 1="A little", 2="Moderately", 3="A lot", 4="Extremely").
  Each domain consists of 6 items. The score is ranging between 0 and 48 and a higher score indicates a worse eating behaviour (greater desire to eat and/or lower capacity to resist).
Absolute change from baseline to Week 76 in glycosylated haemoglobin A1c (HbA1c) (%) | at baseline, at week 76
Absolute change from baseline to Week 76 in HbA1c (mmol/mol) | at baseline, at week 76
Absolute change from baseline to Week 76 in fasting plasma glucose (FPG) (mg/dL) | at baseline, at week 76
Absolute change from baseline to Week 76 in fasting plasma insulin (FPI) (mIU/L) | at baseline, at week 76
Absolute change from baseline to Week 76 in total cholesterol (mg/dL) | at baseline, at week 76
Absolute change from baseline to Week 76 in high density lipoprotein (HDL) (mg/dL) | at baseline, at week 76
Absolute change from baseline to Week 76 in low density lipoprotein (LDL) (mg/dL) | at baseline, at week 76
Absolute change from baseline to Week 76 in very-low-density lipoprotein (VLDL) (mg/dL) | at baseline, at week 76
Absolute change from baseline to Week 76 in triglycerides (mg/dL) | at baseline, at week 76
Absolute change from baseline to Week 76 in free fatty acids (mg/dL) | at baseline, at week 76
Absolute change from baseline to Week 76 in alanine aminotransferase (ALT) (U/L) | at baseline, at week 76
Absolute change from baseline to Week 76 in aspartate aminotransferase (AST) (U/L) | at baseline, at week 76
Relative change from baseline to Week 76 in liver fat content (%), assessed by Magnetic resonance imaging proton density fat fraction (MRI-PDFF) | at baseline, at week 76
Absolute change from baseline to Week 76 in total fat mass (percentage [%]) assessed by MRI for body composition | at baseline, at week 76
Absolute change from baseline to Week 76 in total fat mass (volume [L]) assessed by MRI for body composition | at baseline, at week 76
Absolute change from baseline to Week 76 in lean body mass (percentage [%]) assessed by MRI for body composition | at baseline, at week 76
Absolute change from baseline to Week 76 in lean body mass (volume [L]) assessed by MRI for body composition | at baseline, at week 76
Absolute change from baseline to Week 76 in visceral fat mass (percentage [%]) assessed by MRI for body composition | at baseline, at week 76
Absolute change from baseline to Week 76 in visceral fat mass (volume [L]) assessed by MRI for body composition | at baseline, at week 76
Absolute change from baseline to Week 76 in contractile thigh muscle volume (percentage [%]) assessed by MRI for body composition | at baseline, at week 76
Absolute change from baseline to Week 76 in contractile thigh muscle volume (volume [L]) assessed by MRI for body composition | at baseline, at week 76
Absolute change from baseline to Week 76 in sub-cutaneous fat volume (volume [L]) assessed by MRI for body composition | at baseline, at week 76
Absolute change from baseline to Week 76 in sub-cutaneous fat volume (percentage [%]) assessed by MRI for body composition | at baseline, at week 76

CONTACTS AND LOCATIONS:
Locations (28):
- Japan (28):
  - Hosokawa Surgery Clinic, Aichi, Nagoya
  - Nagoya City University Hospital, Aichi, Nagoya
  - Chiba University Hospital, Chiba, Chiba
  - Gifu University Hospital, Gifu, Gifu
  - Jiyugaoka Yamada Clinic, Hokkaido, Obihiro
  - Yamasaki Family Clinic, Hyogo, Amagasaki
  - Kobe University Hospital, Hyogo, Kobe
  - Motomachi Takatsuka Naika Clinic, Kanagawa, Yokohama
  - Morinagaueno Clinic, Kumamoto, Kumamoto
  - Yoshimura Clinic, Kumamoto, Kumamoto
  - Medical Corporation KEISEIKAI Kajiyama Clinic, Kyoto, Kyoto
  - Ijinkai Takeda General Hospital, Kyoto, Kyoto
  - Osaka Metropolitan University Hospital, Osaka, Osaka
  - OCROM Clinic, Osaka, Suita
  - Saino Clinic, Saitama, Tokorozawa
  - Dojinkinenkai Meiwa Hospital, Tokyo, Chiyoda-ku
  - Suidoubashi Medical Clinic, Tokyo, Chiyoda-ku
  - Tokyo-Eki Center-building Clinic, Tokyo, Chuo-ku
  - Tokyo Center Clinic, Tokyo, Chuo-ku
  - Fukuwa Clinic, Tokyo, Chuo-ku
  - Tokyo Asbo Clinic, Tokyo, Chuo-ku
  - New Medical Research System Clinic, Tokyo, Hachioji
  - Shimamura Kinen Hospital, Tokyo, Nerima-ku
  - Clinical Research Hospital Tokyo, Tokyo, Shinjuku-ku
  - HS Clinic, Tokyo, Shinjuku-ku
  - ToCROM Clinic, Tokyo, Shinjyuku-ku
  - Shinei Medical Healthcare Clinic, Tokyo, Suginami-ku
  - Ikebukuro Metropolitan Clinic, Tokyo, Toshima-ku

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com